CLINICAL TRIAL: NCT03130907
Title: The Role of Ureteral Stenting Following Uncomplicated Ureteroscopy for Ureteral and Renal Stones: A Randomized, Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Antonio Uniformed Services Health Education Consortium (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amy Reed, Principal Investigator, San Antonio Uniformed Services Health Education Consortium
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C.2017.070
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Ureteroscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Stent (Active Comparator)
  Interventions: Device: Placement of ureteral stent
- No stent (Experimental)
  Interventions: Device: Placement of ureteral stent

INTERVENTIONS:
Device: Placement of ureteral stent — will randomize groups to either receive a postoperative ureteral stent or not.

SUMMARY:
It is well established that uncomplicated distal ureteroscopy can be safely performed without leaving a ureteral stent. However, many urologists continue to leave ureteral stents following uncomplicated ureteroscopy, regardless of stone location, due to concerns for post-operative complications, patient symptoms and to reduce unplanned medical visits. There is a paucity of data regarding the utility of stent placement for proximal ureteral or renal stones following ureteroscopy. We have designed a prospective, randomized controlled trial to evaluate the role of ureteral stent placement following ureteroscopy and pyeloscopy in proximal and renal stones.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients age ranges 18-89 with solitary or multiple proximal ureteral or renal stones 1.5cm or smaller measured in the longest dimension on preoperative imaging (CT or xray). Proximal ureteral stones are those proximal to the pelvic brim in the ureter.

Exclusion Criteria:

* Stone size greater than 1.5 cm on preoperative imaging
* Pregnancy
* Stent placement prior to ureteroscopy ("pre-stented patients")
* Patients with solitary kidney

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-05-16 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 30 days
  ED returns, Unplanned OR returns, admissions, UTIs

SECONDARY OUTCOMES:
Subjective patient symptom scores | 6 weeks
  symptom questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- BAMC, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided